CLINICAL TRIAL: NCT01759979
Title: Randomized Trial of Combination of Cholangioscopic Guided Laser Lithotripsy and Conventional Mechanical Versus Conventional Mechanical Methods for the Endoscopic Removal of Large Bile Duct Stones
Brief Title: Laser Versus Mechanical Lithotripsy of Bile Duct Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, James Buxbaum, Director of Endoscopy, Los Angeles County Hospital, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-11-00718
Record Dates: First submitted 2012-12-31; First posted 2013-01-03 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Choledocholithiasis
Keywords: Cholelithiasis, Common Bile Duct; Choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser and mechanical lithotripsy (Experimental): Bile duct stones with be treated with cholangioscopy guided laser therapy in addition to mechanical basket and balloon techniques.
  Interventions: Procedure: Laser and mechanical lithotripsy
- Mechanical lithotripsy (Active Comparator): Patients in the mechanical lithotripsy arm will undergo treatment only with basket and balloon for removal of large stones.
  Interventions: Procedure: Mechanical Lithotripsy

INTERVENTIONS:
Procedure: Laser and mechanical lithotripsy — Patients will undergo cholangioscopy guided laser treatment in addition to treatment with mechanical lithotripsy using basket and balloon techniques.
  Other Names: Spyglass cholangioscopy; Holmium laser lithotripsy
  Arms: Laser and mechanical lithotripsy
Procedure: Mechanical Lithotripsy — Patients in the mechanical lithotripsy arm will undergo treatment only with basket and balloons to facilitate stone removal but not laser lithotripsy.
  Arms: Mechanical lithotripsy

SUMMARY:
Very large bile duct stones are difficult to remove. The prefered method involves an endoscopic procedure known as endoscopic retrograde cholangiopancreatography (ERCP)performed using a special side viewing endoscope. In the past small baskets passed through the scope into the bile duct have been used to remove most stones using mechanical force.

Recently very small scopes known as cholangioscope have been introduced through the side viewing endoscope directly into the bile duct. These cholangioscopes may be used to guide laser therapy of bile duct stones. The investigators suspect that stone destruction using cholangioscopy guided laser stone destruction may enable bile duct stones to be removed more quickly and safely when added to the mechanical techniques.

DETAILED DESCRIPTION:
TITLE: Randomized trial of combination of cholangioscopic guided laser lithotripsy and conventional mechanical versus conventional mechanical methods for the endoscopic removal of large bile duct stones

STUDY ARMS: Laser guided lithotripsy and conventional methods vs conventional methods alone alone

BACKGROUND AND HYPOTHESES: Large bile duct stones are challenging to remove at time of endoscopic retrograde cholangiopancreatography (ERCP) and classically have required the utilization of mechanical baskets and balloons. These maneuvers may be associated with bile duct trauma, bleeding, pancreatitis, and the requirement for additional procedures. Many patients require multiple sessions using conventional mechanical approaches. A recent prospective audit of patients undergoing ERCP during the past year at LAC+USC Medical Center indicates that of approximately 500 procedures more than 250 were for bile duct stones and 100 (40%) required multiple procedures and stent placement. Scheduling challenges and limited resources make it difficult for many of these patients to return for stent changes and increases the risk of complications including cholangitis.

Cholangioscopy enables therapeutic intervention including intracorporeal electro-hydraulic and laser lithotripsy for biliary stone disease with favorable efficacy and safety. Direct visualization by cholangioscopy minimizes the risk of laser related bile duct injury and is potentially much less traumatic and more efficacious than traditional mechanical approaches.

A recent 15 center prospective clinical cohort study demonstrated a high success rate, 89%, and low rate of complications, 7.5%, for the single user cholangioscopy system. In a group of patients who underwent stone removal using the cholangioscope introduced laser or electrohydraulic systems the success even higer 92% and complications potentially lower. Available literature indicates that in cases in which ERCP with mechanical lithotripsy is required the complication rate is approximately 5-12% and risk of cholangitis is 1.4-4%. If ERCP is performed with laser lithotripsy in addition to conventional mechanical methods the complications rate is 6.1% and risk of cholangitis is 2.4%. Cholangioscopy guided laser treatment to enhance stone removal is currently widely used by gastroenterologists at academic centers including the hospitals of the University of Southern California as well as in leading community centers such as the Kaiser Permanente Hospitals of Southern California. While it is a standard of care procedures for large bile duct stones studies directly comparing its efficacy to traditional mechanical approaches are needed.

The long term goal of this project is to assess whether the addition of cholangioscopy guided laser lithotripsy facilitates the removal of large bile duct stones at time of ERCP. Previous prospective studies have demonstrated that the technology is safe and method feasible.

The goal of this pilot study will be to determine the effect size of the difference between laser lithotripsy vs currently available methods on stone removal with the aim of estimating sample size for a fully powered randomized trial. Additional aims will be to assess for procedure duration, cost, and the number of additional procedures required for stone clearance. Complications, hospitalization related to stent dysfunction (frequently placed between lithotripsy sessions), and eventual need for surgery will also be outcomes. Healing time and time prior to return to work will also be outcomes.

OBJECTIVES AND PURPOSE: This is a pilot project to measure the effect of cholangioscopy guided laser lithotripsy in addition to the currently available methods. Large multicenter prospective studies have already demonstrated that the technique is safe and feasible. The overall aims are to assess whether laser lithotripsy combined with conventional methods enhances the rate, efficacy, and cost of stone removal compared to conventional methods including mechanical lithotripsy.

STUDY DESIGN: The study will be a prospective single blind randomized control trial. All patients presenting with choledocholithiasis will be considered for the study. If their ultrasound, computed tomography, and magnetic resonance imaging demonstrates a large stone (>1cm) or biliary dilatation (>1cm) and they do not fulfill the exclusion criterion they will be consented for the study. Randomization will be stratified based on whether or not the procedure is a first or repeat ERCP.

At that point the full time study coordinator will use a computer generated randomization schedule with concealed allocation to generate a 2:1 assignment (laser versus conventional).

At the time of the cholangiogram, which is done immediately prior to stone removal, an assessment will be made by the attending endoscopist to confirm that the stone is greater than 1cm in size.

If confirmed, stone removal will then be attempted using laser lithotripsy using a holmium probe introduced using a single operator cholangioscopy system versus conventional methods. Conventional methods including mechanical baskets and balloon may also be used to remove debris following laser lithotripsy in the laser lithotripsy group. The cholangioscope will not be introduced in those randomized to mechanical lithotripsy and conventional methods alone will be employed. Stents will be placed at the discretion of the attending endoscopist in both groups.

Multiple ERCP procedures may be required to remove the stones. Patients will remain in their assigned treatment groups during subsequent studies. Whether the stones can be successfully removed by the end of the course of therapy and the number of ERCP required for stone clearance are outcomes of interest.

The patients will be blinded to whether or not the cholangioscope was used.

The patient will be followed clinically by the principal investigator assisted by a full time study coordinator daily on the inpatient basis and by a bimonthly phone call on the outpatient basis until 2 months after complete clearance of stones from the bile duct has been confirmed.

DEVICE INFORMATION: The following devices will be used:

Spyglass Direct Visualization System Coherent Holmium Laser VP

Spyglass Direct Visualization System is made by Boston Scientific and the Coherent Holmium Laser VP are produced by Convergent Laser Technologies but is rented by Mobile Med.

All devices used in the study are approved by the FDA for this indication.

SELECTION AND WITHDRAWAL OF SUBJECTS

See Inclusion/Exclusion Criterion

STRATIFICATION/DESCRIPTIVE FACTORS/RANDOMIZATION SCHEME

Patient will be stratified by whether or not they have undergone a prior ERCP or whether the procedure in question is their first ERCP.

The descriptive factors that will be recorded for each patient enrolled in the study include: age, race, gender, and comorbidities at time of presentation.

Following stratification by whether or not they have undergone an ERCP, a computer generated randomized schedule with concealed allocation will generate a 2:1 assignment for the patient, placing them into either the intervention arm (laser lithotripsy using a holmium probe introduced using a single operator cholangioscopy system) or the control arm (conventional methods). As this is a pilot study, designed to gauge the extent of treatment effect and power a larger study 60 patients will be enrolled.

ASSESSMENT OF EFFICACY AND SAFETY

Side effects/Toxicities to be monitored.

Patients in either group may develop post procedure pain, pancreatitis, cholangitis, bile duct injury, or bleeding.

Adverse Event Reporting:

All adverse events will be reported to the principal investigator. The study physicians and coordinator will meet monthly to review these. Adverse events will be reported to the IRB, Data Monitoring Committee, and included in publications.

Data Monitoring Committee:

The study physicians and coordinator will meet monthly to review any adverse events. After no more than 50 patients have been collected all data will be reviewed by a monitoring board including the PI, coinvestigators, study coordinator, and two senior physicians who are part of the clinical gastroentrology faculty

CRITERIA FOR EVALUATION AND ENDPOINT DEFINITIONS

Endpoint Definitions The principle endpoint will be the endoscopic clearance of ductal stones during the course of therapy. Secondary endpoints will be to assess for procedure duration, cost, and the number of procedures required for stone clearance. Complications, hospitalization related to stent dysfunction (frequently placed between lithotripsy sessions), and need for bile duct surgery will also be endpoints.

STATISTICAL CONSIDERATIONS

Descriptive statistics will be performed for all patient characteristics and pre-treatment clinical measures, and comparisons between groups made to ensure balanced. Any variables significantly different between groups will be included in further models as covariates. Intent to treat will be tested for the primary outcome of clearance of ductal strons will be tested using Fisher's exact chi-squared to compare the rate of clearance between groups. Results from this test will allow for estimation of sample size for a fully powered clinical trial. This same method will be used to test dichotomous secondary outcomes: hospitalization related to stent dysfunction and further bile duct surgery. Other secondary aims, which include the count of complications, healing time, and time prior to returning to work will be tested using Poission regression. Total cost will be compared using independent t-tests. Alpha = 0.05 for all analyses. Additionally, because this is a pilot study, effect sizes will be computed to determine potential clinical relevance of outcomes. Statistical analyses will be performed by biostatisticians at the Biostatistical and Bioinformatics Resource Group within the SC CTSI.

ELIGIBILITY:
Inclusion Criteria:

* Bile duct stone >1cm demonstrated on ultrasound, computed tomography, or magnetic resonance imaging
* Bile duct dilatation >1cm

Exclusion Criteria:

* Biliary, gallbladder or pancreatic malignancy
* Pregnant
* Prior biliary diversion surgery
* Under age 18
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Bile Duct Stone Clearance | 12 months
  Confirmation that no further stones remain in the bile duct of the patient by cholangiography. Additionally, serum laboratory abnormalities in AST, ALT, Alkaline Phophatase, or bilirubin, or epigastric abdominal pain attributable to bile duct stones.

SECONDARY OUTCOMES:
Number of ERCP | 12 months
  The number of ERCP procedures required from enrollment in study to complete clearance of bile duct stones.
Total Procedure Time | 12 months
  The total time in minutes for all the ERCP procedures required for stone rumoval.
Estimated Procedure Cost | 12 months
  The cost of patient management for bile duct stones based on the cost of the procedure, hospitalization, and associated costs of complications of cholangitis, pancreatitis, perforation, and bleeding.
Cholangitis | 12 months
  Cholangitis after or between ERCP procedures will be defined as a presentation with epigastric abdominal pain, temperature greater than 38.5 Celsius accompanied by either laboratory abnormalities of the AST, ALT, Alkaline Phosphatase, or Bilirubin or abnormal imaging of the biliary tree on ultrasound,computed tomography scan, or magnetic resonance cholangiopancreatography.
Pancreatitis | 12 months
  Pancreatitis following or between ERCP procedures will be defined as the onset of epigastric abdominal pain and either amylase or lipase greater than 3 times the upper limit of normal or findings on ultrasound, computed tomography scan, or magnetic resonance cholangiopancreatography suggestive of pancreatic inflammation.
Bleeding | 12 months
  Bleeding attributable to stone therapy will be defined as a drop in hemoglobin by more than 1 gm/dl following or between ERCP procedures with no other cause identified on standard clinical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: James L Buxbaum, MD, Principal Investigator — University of Southern California
Locations (1):
- Los Angeles County Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee JG. Diagnosis and management of acute cholangitis. Nat Rev Gastroenterol Hepatol. 2009 Sep;6(9):533-41. doi: 10.1038/nrgastro.2009.126. Epub 2009 Aug 4. PMID 19652653
- [Background] Moon JH, Ko BM, Choi HJ, Hong SJ, Cheon YK, Cho YD, Lee JS, Lee MS, Shim CS. Intraductal balloon-guided direct peroral cholangioscopy with an ultraslim upper endoscope (with videos). Gastrointest Endosc. 2009 Aug;70(2):297-302. doi: 10.1016/j.gie.2008.11.019. Epub 2009 Apr 25. PMID 19394010
- [Background] Kim HI, Moon JH, Choi HJ, Lee JC, Ahn HS, Song AR, Lee TH, Cho YD, Park SH, Kim SJ. Holmium laser lithotripsy under direct peroral cholangioscopy by using an ultra-slim upper endoscope for patients with retained bile duct stones (with video). Gastrointest Endosc. 2011 Nov;74(5):1127-32. doi: 10.1016/j.gie.2011.07.027. Epub 2011 Sep 29. PMID 21963070
- [Background] Chen YK, Parsi MA, Binmoeller KF, Hawes RH, Pleskow DK, Slivka A, Haluszka O, Petersen BT, Sherman S, Deviere J, Meisner S, Stevens PD, Costamagna G, Ponchon T, Peetermans JA, Neuhaus H. Single-operator cholangioscopy in patients requiring evaluation of bile duct disease or therapy of biliary stones (with videos). Gastrointest Endosc. 2011 Oct;74(4):805-14. doi: 10.1016/j.gie.2011.04.016. Epub 2011 Jul 18. PMID 21762903
- [Background] Langman MJ, Constantinopoulos A, Bouchier IA. ABO blood groups, secretor status, and intestinal mucosal concentrations of alkaline phosphatase. Nature. 1968 Mar 2;217(5131):863-5. doi: 10.1038/217863a0. No abstract available. PMID 5641153